CLINICAL TRIAL: NCT02856139
Title: The Director of the Fundus Center of Zhongshan Ophthalmic Center
Brief Title: Appearance of Far Peripheral Retina in Normal Eyes by Ultra-widefield Fluorescein Angiography
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, the Director of the Fundus Center of Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2016036
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Normal Eyes; Peripheral Retina
Keywords: ultra-widefield fluorescein angiography; peripheral retina; normal eyes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 (MB- and VL-): without mottled fluorescent band (MB) and vascular leakage (VL)
- 2 (MB+ and VL-): with mottled fluorescent band (MB), without vascular leakage (VL)
- 3 (MB-/+ and VL+): with or without mottled fluorescent band (MB), with vascular leakage (VL)

SUMMARY:
PURPOSE: To characterize the appearance of the far peripheral retina of normal eyes using ultra-widefield fluorescein angiography (UWFA).

DESIGN: Prospective observational case series. METHODS: This study enrolled normal eyes with best corrected visual acuity ≥ 20/20, refractive error < 3.00D, and without visible retinal pathologic changes under a slit lamp-based condensing lens. The far peripheral retina was detected by UWFA. Ciliary body thickness (CBT) at 3 mm (CBT1) and 2 mm (CBT2) posterior to the scleral spur was measured by ultrasound biomicroscopy.

DETAILED DESCRIPTION:
PURPOSE: To characterize the appearance of the far peripheral retina of normal eyes using ultra-widefield fluorescein angiography (UWFA).

DESIGN: Prospective observational case series. METHODS: This study enrolled normal eyes with best corrected visual acuity ≥ 20/20, refractive error < 3.00D, and without visible retinal pathologic changes under a slit lamp-based condensing lens. Demographic and clinical data such as age, sex, and reasons for undergoing FA were collected. The far peripheral retina was detected by UWFA. The fundal fields obtained using the Heidelberg ultra-widefield lens in a single shot and in montage images were compared with those acquired using the Heidelberg conventional 55° lens. The signs at the peripheral retina detected by UWFA were described and grouped. Ciliary body thickness (CBT) at 3 mm (CBT1) and 2 mm (CBT2) posterior to the scleral spur was measured by ultrasound biomicroscopy.

ELIGIBILITY:
Inclusion Criteria:

* best corrected visual acuity ≥ 20/20
* refractive error < 3.00D
* without visible retinal pathologic changes under a slit lamp-based condensing lens

Exclusion Criteria:

* history of ocular surgery
* presence of ocular or systemic diseases
* opacity of refractive media, which interfered with the peripheral retina image quality

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the fundus outpatient clinic in Zhongshan ophthalmic center who meet the standard of inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Ultra-widefield fluorescein angiography findings at the far peripheral retina of normal eyes | from November 2014 to January 2016

SECONDARY OUTCOMES:
Ciliary body thickness | from November 2014 to January 2016

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No